CLINICAL TRIAL: NCT01438476
Title: Randomized Controlled Trial of Postoperative Thoracic Epidural Analgesia Versus Intravenous Patient Controlled Analgesia (3:1) in Patients Undergoing Liver and/or Pancreatic Resection
Brief Title: Postoperative Thoracic Epidural Analgesia Versus Intravenous Patient-Controlled Analgesia For Liver and/or Pancreas
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0146; NCI-2011-03284 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-09-20; First posted 2011-09-22 (Estimated); Results first posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Liver Cancer; Pancreatic Cancer
Keywords: Liver Cancer; Pancreatic Cancer; Thoracic epidural analgesia; TEA; Intravenous patient-controlled analgesia; IVPCA; Pain control; Quality of life; QOL; Surgical resection
MeSH Terms: conditions — Liver Neoplasms; Pancreatic Neoplasms; Agnosia | interventions — Analgesia, Patient-Controlled; Tea; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IV Pain Management (Experimental): Intravenous analgesia delivered prior to surgery, then patient-controlled following surgical procedures. Hourly post surgery rating level of pain on a scale of 0-10. Questions measure how quickly participant recovers from sedation Day 1 through Day 5 after surgery; approximately 20-40 minutes.
  Interventions: Procedure: Intravenous Patient-Controlled Analgesia (IVPCA); Behavioral: Questionnaires; Behavioral: Pain Assessment
- Epidural Pain Management (Experimental): Thoracic epidurals placed preoperatively in either holding area or in operating room. Hourly post surgery rating level of pain on a scale of 0-10. Questions measure how quickly participant recovers from sedation Day 1 through Day 5 after surgery; approximately 20-40 minutes.
  Interventions: Procedure: Thoracic Epidural Analgesia (TEA); Behavioral: Questionnaires; Behavioral: Pain Assessment

INTERVENTIONS:
Procedure: Intravenous Patient-Controlled Analgesia (IVPCA) — Intravenous analgesia delivered prior to surgery, then patient-controlled following surgical procedures.
  Arms: IV Pain Management
Procedure: Thoracic Epidural Analgesia (TEA) — Thoracic epidurals (needle inserted into the space between the covering of spinal cord and the cord itself) placed preoperatively in either the holding area or in the operating room.
  Arms: Epidural Pain Management
Behavioral: Questionnaires — Questions measure how quickly participant recovers from sedation Day 1 through Day 5 after surgery; approximately 20-40 minutes.
  Other Names: Survey
Behavioral: Pain Assessment — Hourly post surgery rating level of pain on a scale of 0-10.

SUMMARY:
The goal of this clinical research study is to learn if there is a difference in patients' quality of recovery if they receive 1 of 2 standard kinds of pain control treatments after surgery on the liver and/or pancreas. Researchers want to learn which method helps people to recover more completely and more quickly after surgery.

The 2 kinds of pain control are intravenous (IV) pain management and epidural pain management.

DETAILED DESCRIPTION:
Study Groups:

If you agree to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups. For every participant assigned to Group 1, 3 participants will be assigned to Group 2. This means you are 3 times more likely to be assigned to Group 2 than you are to Group 1.

* Group 1 will receive IV pain management.
* Group 2 will receive epidural pain management.

Group 1:

IV pain management will be given through a needle in your arm. This needle will be placed when you are either in the holding area or in the operating room. You will have this needle placed no matter if you take part in this study or not. The needle is used to give drugs and manage fluids during surgery.

After surgery, your doctor will set the limit for the highest dose of pain medication that you can receive at any time, but you will be able to use a hand-held button to adjust your drug according to the level of pain you may be having.

If your pain is not well controlled, the study staff may decide you can be switched to Group 2 if it seems to be in your best interest.

Group 2:

Epidural pain management will be given through a needle inserted into the space between the covering of your spinal cord and the cord itself. This area is full of fluid and is called the epidural region. The needle will be placed before your surgery, either in the holding area or in the operating room by the doctor that gives your anesthesia.

If your epidural does not work, the study staff may decide you can be switched to Group 1 if it seems to be in your best interest.

Both Groups:

During your surgery, you will have a catheter (sterile flexible tube) placed in an artery. This catheter will be used to provide additional fluid and blood support and to monitor you during surgery. Your doctor will explain this procedure to you in more detail, and you will be required to sign a separate consent form.

During surgery, blood (about 1 tablespoon) will be drawn before you receive anesthesia. This blood will be drawn using one of the IV lines that you already have in place for your surgery. This blood will be tested to look for certain proteins called cytokines that may help researchers to understand how your body is responding to pain and how pain is affecting the healing process.

You will be asked to sign a separate consent form that describes the surgery and its risks in detail. The study staff will also tell you about the standard pain medications, how they will be given, and the possible risks.

After Surgery:

After your surgery, you will go to the Post-Anesthesia Care Unit (PACU) for recovery. You will have a physical exam to check your recovery. Your vital signs will also be measured. You will be asked how you are feeling. Your doctor(s) will decide whether you will go from the PACU to the intensive care unit (ICU), overnight recovery suite, or will be moved to a regular post-surgical recovery floor room, where your recovery will be watched.

On Days 1, 3, and 5 after your surgery, blood (about 1 tablespoon) will be drawn for cytokine testing. This blood will be drawn along with the other routine blood work that you will have after your surgery.

If you are in Group 2, a member of the MD Anderson Pain Service will check your epidural site every day to make sure that it is working and that there are no problems with the area around your epidural. A nurse will also check during each shift (about every 8-10 hours) to see how well you are able to move and how the epidural is affecting your feeling in the area it is supposed to be working in.

In both groups, you will be asked to rate your level of pain management on a scale of 0-10. When you first come out of surgery, this pain rating will happen about every hour. Your pain will also be rated about every hour if you are assigned to the surgical ICU. When you get to your room (overnight recovery or surgical floor), it will happen about every 4 hours. You can use your call bell to let a nurse know if your pain is intolerable between the nurses checks.

Questionnaires:

Before your surgery, you will fill out questionnaires about the pain and your quality of life. This should take about 20 minutes to complete.

From the day after surgery (Day 1) through Day 5, you will also be asked to fill out questionnaires about your recovery and any side effects and symptoms you may be having from the pain medication. This will take about 20-40 minutes.

While you are in the hospital, you will be asked to answer some questions that will measure how quickly you recover from the sedation used during your surgery. Each shift (about every 8-10 hours), a nurse will ask you questions to find out how quickly you are recovering from anesthesia.

Length of Study Participation:

The pain medication or epidural insertion will be stopped early if you are having intolerable side effects or if the medication is not working.

Your participation in the study will be over after Day 5.

This is an investigational study. IV pain management and epidural pain management are FDA approved and commercially available. Randomly assigning you to a type of pain management and comparing the treatments is being done for research purposes only.

Up to 200 patients will be enrolled in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing liver and/or pancreatic surgical resection for malignancy at MD Anderson Cancer Center.
2. Patients 18 years of age and older. There will be no upper age restriction.
3. Patients must sign a study-specific consent form.
4. Adequate coagulation function within 30 days of surgery: Platelets >/= 100,000/ml; international normalized ratio (INR) </= 1.5; activated partial thromboplastin time (aPTT) </= 40.
5. Patients must have no fever or evidence of infection or other coexisting medical condition that would preclude epidural placement.

Exclusion Criteria:

1. Evidence of severe uncontrolled systemic disease or other comorbidity that precludes liver or pancreatic surgery.
2. History of chronic pain, long-term narcotic use or being considered for chronic pain consultation postoperatively.
3. Anaphylaxis to local anesthetics or narcotics.
4. Previous or current neurologic disease affecting the lower hemithorax or below.
5. Major open abdominal/thoracic surgery in the previous 30 days under general anesthesia, except for total intravenous anesthesia (TIVA).
6. Technical contraindications to epidural placement: previous thoracic spinal surgery or local skin or soft tissue infection at proposed site for epidural insertion.
7. Ongoing use or planned peri-operative use of anticoagulants (not including deep vein thrombosis (DVT) prophylaxis).
8. Known bleeding diathesis or coagulopathy.
9. Educational, psychiatric (untreated or poorly controlled schizophrenia, major depression, or bipolar disorder), or communication (language) barrier that would preclude accurate assessment of postoperative pain and/or ability to answer questionnaires (need to be able to read, comprehend, and answer questions).
10. Inability to comply with study and/or follow-up procedures.
11. Patient refusal to participate in randomization.
12. Pregnant women are excluded from this study; women of childbearing potential (defined as those who have not undergone a hysterectomy or who have not been postmenopausal for at least 12 consecutive months) must agree to practice adequate contraception and to refrain from breast-feeding, as specified in the informed consent.
13. Patients with obvious unresectable disease prior to signing informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2012-01-26 (Actual); Primary Completion 2017-10-18 (Actual); Study Completion 2017-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Nicolas Vauthey, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Cata JP, Velasquez JF, Ramirez MF, Vauthey JN, Gottumukkala V, Conrad C, Kim BJ, Aloia T. Inflammation and pro-resolution inflammation after hepatobiliary surgery. World J Surg Oncol. 2017 Aug 10;15(1):152. doi: 10.1186/s12957-017-1220-6. PMID 28807031
- [Derived] Aloia TA, Kim BJ, Segraves-Chun YS, Cata JP, Truty MJ, Shi Q, Holmes A, Soliz JM, Popat KU, Rahlfs TF, Lee JE, Wang XS, Morris JS, Gottumukkala VNR, Vauthey JN. A Randomized Controlled Trial of Postoperative Thoracic Epidural Analgesia Versus Intravenous Patient-controlled Analgesia After Major Hepatopancreatobiliary Surgery. Ann Surg. 2017 Sep;266(3):545-554. doi: 10.1097/SLA.0000000000002386. PMID 28746153
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During the study period, 178 screened patients were initially eligible for inclusion to the randomized controlled trial.
Pre-assignment Details: Among the 178 eligible patients, 38 patients were excluded due to withdrawal of consent, development of exclusion criteria and/or the finding of unresectable disease at surgery. The study concluded with 140 patients eligible for analysis, with 106 patients allocated to the TEA group and 34 patients allocated to the IV-PCA group.
Groups:
- TEA (Thoracic Epidural Analgesia): Thoracic Epidural Analgesia-TEA Thoracic epidurals placed preoperatively in either holding area or in operating room. Hourly post surgery rating level of pain on a scale of 0-10. Questions measure how quickly participant recovers from sedation Day 1 through Day 5 after surgery; approximately 20-40 minutes.
  Thoracic Epidural Analgesia (TEA): Thoracic epidurals (needle inserted into the space between the covering of spinal cord and the cord itself) placed preoperatively in either the holding area or in the operating room.
  Questionnaires: Questions measure how quickly participant recovers from sedation Day 1 through Day 5 after surgery; approximately 20-40 minutes.
  Pain Assessment: Hourly post surgery rating level of pain on a scale of 0-10.
- IV-PCA (Intravenous Patient-controlled Analgesia): Intravenous Patient-controlled Analgesia IV-PCA: Intravenous analgesia delivered prior to surgery, then patient-controlled following surgical procedures. Hourly post surgery rating level of pain on a scale of 0-10. Questions measure how quickly participant recovers from sedation Day 1 through Day 5 after surgery; approximately 20-40 minutes.
  Intravenous Patient-Controlled Analgesia (IVPCA): Intravenous analgesia delivered prior to surgery, then patient-controlled following surgical procedures.
  Questionnaires: Questions measure how quickly participant recovers from sedation Day 1 through Day 5 after surgery; approximately 20-40 minutes.
  Pain Assessment: Hourly post surgery rating level of pain on a scale of 0-10.
Period: Overall Study
Arm/Group | TEA (Thoracic Epidural Analgesia) | IV-PCA (Intravenous Patient-controlled Analgesia)
Started | 116 | 45
Completed | 106 | 34
Not Completed | 10 | 11
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — No Surgery- Disease | 8 | 10
Not completed — Communication barrier | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TEA (Thoracic Epidural Analgesia) | IV-PCA (Intravenous Patient-controlled Analgesia) | Total
Number analyzed (Participants) | 106 | 34 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 85 | 27 | 112
  >=65 years | 21 | 7 | 28
Age, Continuous [Median (Full Range); unit: years] | 56.3 [48.9 to 62.8] | 57.4 [54.6 to 63.8] | 56.8 [48.9 to 63.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 19 | 62
  Male | 63 | 15 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 2 | 10
  Not Hispanic or Latino | 98 | 32 | 130
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 3 | 14
  White | 89 | 30 | 119
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 106 | 34 | 140
Major hepatectomy [Count of Participants; unit: Participants] | 70 | 20 | 90

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain Experience
Description: The Area Under the Curve (AUC) pain score during the first 48 hours after surgery. Post operative pain was measured during the first 48 hours per unit acuity guidelines. Typically this was at a minimum of every four hours yielding an average number of measures during the first 48 hours. The scale is 0-480 low scores are better.
Time Frame: First 48 hours after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale* hour
Arm/Group | TEA (Thoracic Epidural Analgesia) | IV-PCA (Intravenous Patient-controlled Analgesia)
Number analyzed (Participants) | 106 | 34
score on a scale* hour | 78.6 [49.6 to 115.3] | 105.2 [64.2 to 144.2]

ADVERSE EVENTS:
Time Frame: Patients were assessed during their inpatient hospitalization average and range of length of stay for each arm is provided in the data table.
Arm/Group | TEA (Thoracic Epidural Analgesia) | IV-PCA (Intravenous Patient-controlled Analgesia)
All-Cause Mortality (participants affected / at risk) | 0/106 | 0/34
Serious Adverse Events (participants affected / at risk) | 21/106 | 3/34
Other Adverse Events (participants affected / at risk) | 0/106 | 0/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TEA (Thoracic Epidural Analgesia) (N=106) | IV-PCA (Intravenous Patient-controlled Analgesia) (N=34)
Analgesia (Gastrointestinal disorders) | 13 | 1
Ileus (Gastrointestinal disorders) | 8 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-12): https://cdn.clinicaltrials.gov/large-docs/76/NCT01438476/Prot_SAP_000.pdf